CLINICAL TRIAL: NCT04905706
Title: Three-dimensional Laparoscopic Adrenalectomies for Benign and Malignant Adrenal Tumors
Brief Title: 3D Laparoscopic Adrenalectomies for Adrenal Tumors
Status: Recruiting | Type: Observational
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, José Ignacio Rodríguez-Hermosa, MD, PhD, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Other Study IDs: 2020.141
Record Dates: First submitted 2021-05-14; First posted 2021-05-28 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Adrenal Tumor; Adrenalectomy; Status
Keywords: Three-dimensional laparoscopy; Adrenal tumors; 3D laparoscopic adrenalectomy
MeSH Terms: conditions — Adrenal Gland Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 3D laparoscopic adrenalectomy: Operations are done with an high definition 3D laparoscopic system (Olympus, Tokyo, Japan); all personnel wear polarized glasses to achieve stereoscopic imaging in the operating room. Dissection is realized using a hybrid energy system (Thunderbeat, Olympus Europe Se & Co, Hamburg, Germany).

SUMMARY:
The main drawbacks of conventional 2D laparoscopy are limited depth perception and loss of spatial orientation. High-quality 3D laparoscopy systems might improve surgical outcomes for adrenalectomy.

DETAILED DESCRIPTION:
Over recent decades, technological advances such as improved video imaging (high-definition cameras), better instrumentation for dissection and hemostasis, articulating staplers, and optimized operating room lighting have added safety, efficacy, and precision to minimally invasive procedures. However, until recently, laparoscopy required surgeons to operate in a three-dimensional (3D) space with only two-dimensional (2D) images to guide their movements, resulting in a lack of depth perception and loss of spatial orientation that increased the risk of errors, fatigue, operative time, and operating room stress and made the technique difficult to learn.

High-quality 3D laparoscopy was developed as an alternative to conventional 2D laparoscopy. Several clinical trials and observational studies have compared surgical outcomes between 2D and 3D laparoscopic systems; however, few clinical studies have examined the usefulness of 3D laparoscopy systems for adrenalectomies.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age ≥ 18 years)
* Patients diagnosed with adrenal masses (benign and malignant tumors)
* Underwent a unilateral 3D laparoscopic adrenalectomy from January 2013 to December 2033.

Exclusion Criteria:

* Emergency surgery.
* Open adrenalectomy.
* Bilateral adrenalectomies (open or laparoscopy).
* Patients who underwent laparoscopic adrenalectomy together with another laparoscopic surgical procedure in the same intervention.
* Patients without complete follow-up for at least 30 days after hospital discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (age ≥ 18 years) who underwent a unilateral 3D laparoscopic adrenalectomy for adrenal masses (benign and malignant tumors) from January 2013 to December 2033.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2033-11-30 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications rate of 3D laparoscopic adrenalectomy | Within 30 days after surgery
  Rate of medical and surgical complications within 30 days after surgery using the Dindo-Clavien classification, described as:
  Grade I = Any deviation from the normal postoperative course. Grade 2 = Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Grade III = Requiring surgical, endoscopic or radiological intervention, not under (Grade IIIa) or under general anesthesia (Grade IIIb) Grade IV = Life-threatening complication with single organ (Grade IVa) or Multiorgan dysfunction (Grade IVb) Grade V = Death of a patient.
Length of hospital stay | Up to 4 weeks
  Total length of hospital stay will be recorded in days beginning at admission for surgery until discharge (number of days) .

SECONDARY OUTCOMES:
Conversion rate trough 3D laparoscopic adrenalectomy | Intraoperatively
  Conversion to open surgery (Yes vs No).
Intraoperative bleeding during 3D laparoscopic adrenalectomy | Intraoperatively
  Blood loss during surgery (millilitres)
Operative time trough 3D laparoscopic adrenalectomy | Intraoperatively
  Duration of intervention (minutes)
Routine use of abdominal drainage in 3D laparoscopic adrenalectomy | Intraoperatively
  Use of abdominal drainage intraoperatively (Yes vs No).
Comparison of morbidity between obese and non obese patients operated by 3D laparoscopic system | Within 30 days after surgery
  No obese: <30 kg/m2 Obese: ≥30 kg/m2
Comparison of morbidity in patients with prior abdominal surgery versus non operated by 3D laparoscopic system | Within 30 days after surgery
  Prior abdominal surgery (Yes vs No).
Comparison of morbidity between elderly and young patients operated by 3D laparoscopic system | Within 30 days after surgery
  Young <65 years, Elderly ≥65 years
Comparison of morbidity between American Society of Anesthesiologists I+II and III+IV operated by 3D laparoscopic system | Within 30 days after surgery
  ASA I A normal healthy patient ASA II A patient with mild systemic disease ASA III A patient with severe systemic disease ASA IV A patient with severe systemic disease that is a constant threat to life ASA V A moribund patient who is not expected to survive without the operation ASA VI A declared brain-dead patient whose organs are being removed for donor purposes
Comparison of morbidity between adrenal mass size <6 cm versus ≥6 cm operated by 3D laparoscopic system | Within 30 days after surgery
  Adrenal mass <6 cm, Adrenal mass ≥6 cm
Comparison of adrenal mass diagnosis operated by 3D laparoscopic system | Within 30 days after surgery
  Incidentaloma, Aldosteronoma, Pheochromocytoma, Cushing's Adenoma and malignant adrenal tumors (primary or metastasis)
Comparison of adrenal mass laterality operated by 3D laparoscopic system | Within 30 days after surgery
  Right adrenal mass, left adrenal mass
Comparison of morbidity between 2D versus 3D laparoscopic system | Within 30 days after surgery
  Conversion (Yes vs No), operative time (min), bleeding (ml), Clavien-Dindo Classification

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Dr. Josep Trueta de Girona, Girona, Girona, Spain